CLINICAL TRIAL: NCT03013088
Title: A First in Man Study to Assess the Soundbite Crossing System When Used to Cross Infrainguinal Chronic Total Occlusions
Brief Title: Soundbite Crossing System Peripheral First in Man
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SoundBite Medical Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-PER-2015-01
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Peripheral Artery Disease
Keywords: Chronic; Occlusion; CTO
MeSH Terms: conditions — Peripheral Arterial Disease; Bronchiolitis Obliterans Syndrome; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CTO Crossing (Experimental): With confirmation that the target vessel is completely occluded by the target CTO lesion, the operator shall initially attempt crossing the proximal end of the target CTO lesion by advancing ShockWireTM device ≥ 1cm. The SoundBite Crossing device can be activated as needed to perform the procedure and may be used for the entire length of the lesion(s).
  Interventions: Device: CTO Crossing

INTERVENTIONS:
Device: CTO Crossing — With confirmation that the target vessel is completely occluded by the target CTO lesion, the operator shall initially attempt crossing the proximal end of the target CTO lesion by advancing ShockWireTM device ≥ 1cm. The SoundBite Crossing device can be activated as needed to perform the procedure and may be used for the entire length of the lesion(s).

SUMMARY:
This is a clinical study aimed at demonstrating the safety and product performance of the SoundBite Crossing System. The study shall demonstrate that the SoundBite Crossing System can facilitate passage of a standard guidewire through a Chronic Total Occlusion (CTO) located in the lower extremity arteries without major adverse events related to SoundBite device utilization.

DETAILED DESCRIPTION:
Prospective, multi-center, single-arm, two-phase clinical study. This study will be conducted in two phases.

The first phase will consist of ten (10) subjects enrolled and treated using the SoundBite Crossing System with 30 day follow-up. An analysis shall be performed after 10 subjects undergo treatment with the SoundBite Crossing System and complete 30 day follow-up. This analysis shall be utilized to provide insight into product performance and safety.

The second phase will consist of up to forty (40) subjects enrolled and treated using the SoundBite Crossing System with 30 day follow-up. An analysis will be generated on this subject cohort after 30 day follow-up is complete.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic target leg ischemia, requiring treatment of an infrainguinal artery.
2. Rutherford Category of 2-5.
3. ≥ 18 years of age.
4. Life expectancy > 1 year.
5. Able and willing to provide written informed consent prior to study procedure.
6. Evidence that the target CTO lesion is a de novo or restenotic chronic total occlusion in the SFA (starting at least 1cm distal to the origin of the SFA) and/or popliteal artery (ending at least 1cm proximal to the popliteal trifurcation), confirmed by angiography; AND/OR Evidence that the target CTO lesion is a de novo or restenotic chronic total occlusion and is located below the popliteal trifurcation in the anterior tibial, posterior tibial or peroneal arteries (at least 1 cm distal to the vessel origin, and ending at least 1cm proximal to the dorsalis pedis or plantar arteries), confirmed by angiography.
7. Target CTO lesion is 100% occluded by visual estimate.
8. Target limb has at least one patent (<50% stenosis) tibio-peroneal run-off vessel to the foot confirmed by baseline angiography or magnetic resonance angiography (MRA) or computed tomography angiography (CTA).
9. Target CTO lesion has a cumulative lesion length of no more than 40 cm and terminates at least 1 cm above the ankle or tibio-talar joint.
10. Reference vessel diameter, by visual estimate, is ≥ 4 mm for femoral-popliteal arteries, or ≥ 2 mm for tibial or peroneal arteries.

Exclusion Criteria:

1. History of previous peripheral bypass or stent placement, affecting the target CTO lesion (i.e. target CTO lesion (de novo or restenotic) must be at least 1cm proximal or distal to a surgical bypass graft anastomosis or stent edge to be eligible for treatment).
2. History of receiving a kidney transplant.
3. Current significant acute or chronic kidney disease with a creatinine level > 220 micromoles/Land/or requiring dialysis.
4. Known or suspected active infection at the time of the index procedure, excluding an infection of a lower extremity wound of the target limb.
5. History of an endovascular procedure or open vascular surgery on the index limb within the 30 days prior to enrollment.
6. Any planned surgical or interventional procedure within 30 days after the index procedure.
7. Unstable coronary artery disease or other uncontrolled comorbidity.
8. Myocardial infarction or stroke within 3 months prior to enrollment.
9. Currently pregnant or breast-feeding.
10. Participating in any study of an investigational device, medication, biologic, or other agent within 30 days prior to enrollment that is either a cardiovascular study or could, in the judgement of the Investigator, affect the results of this study.
11. Known significant stenosis or occlusion of inflow tract (upstream disease) not successfully treated before index procedure.
12. Contraindication to antiplatelet medications, anticoagulant medication, or thrombolytic therapy.
13. Current uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/microliter, known coagulopathy, or INR >1.5.
14. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
15. History of heparin-induced thrombocytopenia (HIT).
16. Received thrombolytic therapy within two weeks of enrollment.
17. Known psychiatric disorder which in the judgement of the Investigator could interfere with provision of informed consent, completion of tests, therapy, or follow-up.
18. Clinical/angiographic complication (other than non-flow limiting dissections) attributed to a currently marketed device prior to introduction of SoundBite Crossing System.
19. Acute or sub-acute intraluminal thrombus within the target vessel.
20. Aneurysm (at least twice the reference vessel diameter) located in the target vessel or popliteal artery.
21. Perforation, dissection or other injury of the access or target vessel requiring stenting or surgical intervention.
22. Clinical/angiographic evidence of distal embolization in the target limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Device Success | 30 Day follow-up
  Device Success is the primary endpoint for the study. Device Success is defined as the achievement of Technical Success with freedom from Major Adverse Events through 30 day follow-up, per Independent Physician Reviewer (IPR) adjudication.

SECONDARY OUTCOMES:
Technical Success | At the time of the index procedure
  Technical Success: the ability of the SoundBite Crossing System to facilitate crossing of a target CTO lesion, defined as: The ShockWireTM being advanced by 1cm or more into proximal aspect of target CTO lesion based on angiography; AND Either the ShockWireTM or other commercially available device (e.g. guidewire) is able to cross target CTO lesion.
  Technical Success shall be assessed at the time of the index procedure after all ShockWireTM devices have been used on the target CTO lesion (if more than one ShockWireTM device was utilized to address the target CTO lesion).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Benko, MD, Principal Investigator — CHUS - Centre Hospitalier Universitaire de Sherbrooke - Fleurimont
Locations (2):
- Canada (2):
  - CHUM - Centre Hospitalier de l'Université de Montreal - Hôtel-Dieu, Montreal, Quebec
  - CHUS - Centre Hospitalier Universitaire de Sherbrooke - Freurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No